CLINICAL TRIAL: NCT01331746
Title: Randomised, Double-blind, Placebo-controlled Phase II Proof-of-concept Study of APD515 Solution for Oromucosal and Oral Administration for Relief of Xerostomia in Patients With Cancer
Brief Title: Proof-of-concept (PoC) Study of APD515
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DX10008
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Xerostomia in Advanced Cancer Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- APD515 (Experimental): Active APD515 treatment 20 mg qds for 7 days
  Interventions: Drug: APD515
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD515 — 20 mg oromucosal-oral administration qds for 7 days
  Arms: APD515
Drug: Placebo — qds for 7 days
  Arms: Placebo

SUMMARY:
A study to look at the effectiveness of a drug called APD515, designed to be applied to the lining inside the mouth, at relieving dryness of the mouth. Study will compare one week of treatment with APD515 to one week of treatment with matching placebo to see which has better effect on patient's mouth dryness, according to their own score.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Able and willing to give written informed consent.
* Confirmed primary neoplasm at any site (apart from non-melanoma skin cancers), for which first-line cytotoxic therapy has been completed more than one month prior to study entry. Ongoing palliative, hormonal, cytostatic or "targeted" (e.g., monoclonal antibody, tyrosine kinase inhibitor, etc) therapy is permitted, provided that the risk of oral mucositis in the subject is not judged to be significant.
* Subjective complaint of dry mouth, ongoing for at least two weeks prior to study entry.
* Capacity for salivary stimulation, as demonstrated by stimulated whole saliva flow rate > unstimulated whole saliva flow rate.
* Karnofsky performance score ≥ 60% or ECOG performance status ≤ 2.
* Adequate renal and hepatic function and hydration status:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5 * upper limit normal (ULN);
  * Serum urea < 1.5 * ULN and serum urea:creatinine ratio < 100 (where urea and creatinine expressed in the same units);
  * Plasma sodium ≤ ULN.
* Adequate haematological function:

  * Haemoglobin ≥ 9 g/dL;
  * White blood count ≥ 1.0 * 10^9/L;
  * Platelet count ≥ 50 *x 10^9/L.
* For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (e.g., abstinence from sexual intercourse, surgical sterilisation (of subject or partner) or a double-barrier method of contraception such as either an intra-uterine device (IUD) or an occlusive cap with spermicide, in conjunction with partner's use of a condom) during the study and for a period of at least 48 hours afterwards.

Exclusion Criteria:

* Confirmed diagnosis of Sjögren's syndrome.
* Prior radiotherapy for head & neck cancer, or other substantial doses of radiation delivered to the area of the mouth or salivary glands.
* Significant, symptomatic disease of the oral cavity, including oral candidosis or oral mucositis.
* Allergy to active ingredient or any of the excipients of APD515.
* Use of oral or topical (including ocular) pilocarpine or cevimeline in the two weeks prior to enrolment.
* Concomitant use of procainamide, quinidine or ganglionic blocking agents such as mecamylamine, pentolinium and trimethaphan.
* Intestinal or urinary obstruction.
* Myocardial infarction or intestinal anastomosis within the previous 6 months.
* Participation in an investigational drug or device study within 1 month prior to study entry.
* For female subjects only, a positive pregnancy test.
* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Xerostomia score | 1 week
  Change in score on 100 mm visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MD, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (11):
- Denmark (3):
  - Århus University Hospital, Aarhus
  - University of Copenhagen, Copenhagen
  - Hillerød Hospital, Hillerød
- United Kingdom (8):
  - Sue Ryder Leckhampton Court Hospice, Cheltenham
  - Coventry and Warwickshire Partnership Trust, Coventry
  - Royal Surrey County Hospital, Guildford
  - John Eastwood Hospice, Mansfield
  - Priscilla Bacon Lodge, Norwich
  - City Hospital Hayward House Specialist Palliative Care Unit, Nottingham
  - Scarborough General Hospital, Scarborough
  - Severn Hospice, Shrewsbury